CLINICAL TRIAL: NCT06799234
Title: Phase 2 Trial to Assess the Immunogenicity and Safety of the ChAdOx1 RVF Vaccine Against Rift Valley Fever in Adults in Kenya
Brief Title: Safety and Immunogenicity of a Candidate Rift Valley Fever Vaccine (RVF003)
Acronym: RVF003
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OxTREC 3/24; KEMRI/SERU/CGMRC/314/4960 (Other: Kenya Medical Research Institute); PACTR202406789723926 (Registry Identifier: Pan African Clinical Trial Registry); PPB/ECCT/24/07/03 (Other: Kenya Pharmacy and Poisons Board)
Record Dates: First submitted 2024-09-20; First posted 2025-01-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Rift Valley Fever
MeSH Terms: conditions — Rift Valley Fever | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blinded phase 2 trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants will be blinded to the allocations. Only the pharmacist and the nurse administering the vaccine will be unblinded. The allocation will be to one of the three treatment arms per a computer-generated randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single dose ChAdOx1 RVF (Experimental): Group 1, composed of 120 participants, will receive a single dose of ChAdOx1 RVF vaccine at baseline and a single dose of rabies vaccine 3 months later
  Interventions: Biological: ChAdOx1 RVF; Biological: Rabies Vaccine
- Double dose ChAdOx1 RVF (Experimental): Group 2, composed of 60 adults, will receive two doses of ChAdOx1 RVF; the first dose at baseline and the second dose 3 months later.
  Interventions: Biological: ChAdOx1 RVF
- Rabies vaccine (Active Comparator): Group 3, composed of 60 adults, will receive two doses of rabies vaccine; the first dose at baseline and the second dose 3 months later
  Interventions: Biological: Rabies Vaccine

INTERVENTIONS:
Biological: ChAdOx1 RVF — One 0.36mL dose contains 5x10^10vp ChAdOx1 RVF.
  Arms: Double dose ChAdOx1 RVF; Single dose ChAdOx1 RVF
Biological: Rabies Vaccine — 1mL per dose
  Arms: Rabies vaccine; Single dose ChAdOx1 RVF

SUMMARY:
The goal of this clinical trial is to learn if ChAdOx1 RVF, a candidate vaccine against RVF, provides an adequate immune response and determine its safety among Kenyan adults. The main aims are:

* To assess the proportion of individuals mounting an immune response following vaccination with a single dose of ChAdOx1 RVF
* To monitor occurrence of any adverse events following vaccination
* To assess whether two doses of ChAdOx1 RVF elicit an immune response that is more durable than that generated by a single dose of ChAdOx1 RVF

Researchers will compare ChAdOx1 RVF vaccine to a rabies vaccine in 240 participants. Participants will be randomly allocated to one of three study groups and vaccinated with ChAdOx1 RVF or a control Rabies vaccine as follows.

Group 1, composed of 120 participants, will receive a single dose of ChAdOx1 RVF vaccine at baseline and a single dose of rabies vaccine 3 months later. Group 2, composed of 60 adults, will receive two doses of ChAdOx1 RVF; the first dose at baseline and the second dose 3 months later. Group 3, composed of 60 adults, will receive two doses of rabies vaccine; the first dose at baseline and the second dose 3 months later.

Participants will receive daily phone calls after each vaccination for the following six days to gather information on any symptoms they may experience. Participants will be instructed to contact the study team at any time should they experience any clinical symptoms. Blood samples will be collected at baseline (before vaccination) and at scheduled follow-up visits (8 visits over the duration of the study, i.e. days 7, 14, 28, 84, 91, 112, 365 and 540 after the first vaccination) for monitoring of immune responses. Up to 20mls of blood will be collected at each scheduled visit. Participants will be followed-up for 18 months from the first dose of vaccine.

Adverse events following vaccination will be monitored throughout the study and reviewed by an independent Data and Safety Monitoring Board (DSMB)

DETAILED DESCRIPTION:
Rift Valley fever (RVF) is a mosquito-borne viral illness that was first discovered in Kenya in 1930 and is now present in many parts of the country including Kilifi and other coastal counties. The disease primarily affects humans and livestock (sheep, goats, cattle) and has spread throughout much of Africa and part of the Middle East. In humans, RVF is characterized by a wide range of symptoms ranging from self-limiting febrile illness to life-threatening bleeding complications and miscarriage in pregnant women. Overall mortality from RVF is thought to be <1%; however, case fatality rates among patients with bleeding complications can be as high as 50% and other serious outcomes of disease such as blindness can occur with some forms of the disease. In livestock, more than 90% of young animals affected by RVF die and spontaneous abortion in almost all pregnant animals on a farm is typical. Vaccines against RVF are available for livestock, but no licensed vaccines are currently available for human use. Owing to the potential for a public health emergency arising from RVF epidemics, both the World Health Organization (WHO) and the African Union have identified the development of a human RVF vaccine as an urgent priority.

The aim of the trial is to answer the question of whether ChAdOx1 RVF, a candidate vaccine against RVF, provides an adequate immune response and determine its safety among Kenyan adults. The vaccine has been found to be safe, able to generate a strong durable immune response, and to confer protection against RVF in all major livestock species affected by the disease. In human phase 1 trials in adults in the United Kingdom and Uganda, a single dose of ChAdOx1 RVF was also shown to be safe and able to generate a strong immune response. Further evaluation of ChAdOx1 RVF in larger populations in areas where RVF epidemics occur is necessary for subsequent licensure and deployment of the vaccine. This study will evaluate the safety of, and immune response generated by ChAdOx1 RVF vaccine in adults in Kenya. The main aim is to assess the proportion of individuals mounting an immune response following vaccination with a single dose of ChAdOx1 RVF, and occurrence of any adverse events following vaccination. A secondary aim of the study is to assess whether two doses of ChAdOx1 RVF elicit an immune response that is more durable than that generated by a single dose of ChAdOx1 RVF.

This phase 2 vaccine trial will be conducted among adults aged 18-50 years resident within the Kilifi Health and Demographic Surveillance System (KHDSS) in Kilifi County, Kenya where RVF outbreaks have previously occurred. A total of 240 enrolled adults will be randomly allocated for vaccination with ChAdOx1 RVF or with rabies vaccine as a control.

Prior to enrolment, study participants will complete screening procedures to ensure they are in good health after they have given written informed consent. Participants will be screened for any significant health problems. This will include sampling of blood and urine for a series of tests to ensure eligibility. volunteers found eligible to participate will be randomly allocated to one of three study groups and vaccinated with ChAdOx1 RVF or a control Rabies vaccine as follows. Group 1, composed of 120 participants, will receive a single dose of ChAdOx1 RVF vaccine at baseline and a single dose of rabies vaccine 3 months later. Group 2, composed of 60 adults, will receive two doses of ChAdOx1 RVF; the first dose at baseline and the second dose 3 months later. Group 3, composed of 60 adults, will receive two doses of rabies vaccine; the first dose at baseline and the second dose 3 months later. All screening procedures, sampling and vaccination will be done at the study clinic within the KEMRI-Wellcome Trust Research Programme. The choice of Rabies vaccine as a control is due to its good safety profile and the benefit that rabies vaccination offers participants given the risk of rabies in Kenya. After each vaccination, participants will receive daily phone calls for the following six days to gather information on any symptoms they may experience. Participants will be instructed to contact the study team at any time should they experience any clinical symptoms. Blood samples will be collected at baseline (before vaccination) and at scheduled follow-up visits (8 visits over the duration of the study, i.e. days 7, 14, 28, 84, 91, 112, 365 and 540 after the first vaccination) for monitoring of immune responses. Up to 20mls of blood will be collected at each scheduled visit. Participants will be followed-up for 18 months from the first dose of vaccine. Adverse events following vaccination will be monitored throughout the study and reviewed by an independent Data and Safety Monitoring Board (DSMB).

Participants will benefit by knowledge of their general health status; they will also have close oversight and treatment support from the study team although this will primarily be for risk monitoring. All participants will also be offered the opportunity to receive a complete course of the rabies vaccine at the end of the study. During vaccination and when collecting blood samples, the participants may experience some discomfort, pain and occasionally, bruising at the injection site, which gets better after a short while. With any vaccination there is a risk of rare serious adverse events, such as a severe allergic reaction. In case of this unlikely event, medication for treating allergic reactions is kept in the clinic room and the investigators are appropriately trained in the management of allergic reactions. An extremely rare but serious blood clot condition that can lead to death or serious long-term disability has been observed among individuals vaccinated with a COVID-19 vaccines made using the technology used to make the ChAdOx1 RVF vaccine. A very rare condition that affects the nervous system, called Guillain-Barre Syndrome, has also been observed with COVID-19 vaccines. However, it is not clear whether other vaccines made with the ChAdOx1 technology will carry a similar risk of inducing the clotting condition or the nervous system condition. All participants will be provided with this information via the informed consent form and will be kept updated should further information become available. Participants will be specifically counselled on symptoms that could be warning signs of serious clotting events, and any cases managed as per local Ministry of Health guidelines. Participants will be compensated for study-related out-of-pocket expenses for each clinic study visit, reimbursed for transport costs incurred, and pay for their costs of hospitalization in a government facility for any new illness that develop during the study period.

If found to be safe and good in generating protective immune responses, the ChAdOx1 RVF vaccine will be developed further and licensed for use in controlling RVF in humans. The study will start upon receipt of ethical and regulatory approvals. The estimated trial period, starting from when the first participant is screened for eligibility to when the final participant has had their last follow-up visit and the trial database is locked, will be 24 months. The total study duration including the time taken to obtain ethics and regulatory approvals, community engagement activities and post-study reporting to take approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-50 years
* For females only, willingness to practice continuous effective contraception up to one month following the second vaccination (i.e. duration of 4 months starting from enrolment) and a negative pregnancy test on the day(s) of screening. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include combined oral contraceptives, injectable progestogen, implants of etenogestrel or levonorgestrel, intrauterine device. Female participants will be asked for written confirmation of any family planning methods used by provision of health records. These records will be reviewed and counselling for adherence done at each study visit as per the protocol schedule of attendances. Participants who do not have adequate methods of contraception will be referred to their local dispensary where this will be dispensed for free or to Kilifi County Hospital (KCH). Costs incurred for obtaining contraception at KCH will be covered by the study.
* Agreement to refrain from blood donation during the course of the study
* Able and willing to provide written informed consent
* Plan to remain resident in the study area for 18 months following vaccination

Exclusion Criteria:

* Prior receipt of any vaccines (licensed or investigational) ≤30 days before enrolment and/or planned receipt of a vaccine ≤30 days after enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week (e.g., more than 2 bottles of 500mls Tusker (beer) a day, more than 2 large glasses of 12% wine per day)
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (HCV)
* Prior natural exposure to RVFV as determined by seropositivity for RVFV antigens by ELISA
* Any clinically significant abnormal finding on screening biochemistry, hematology or coagulation blood tests or urinalysis
* Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the participant because of participation in the study, affect the ability of the individual to participate in the study or impair interpretation of the study data
* History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), history of antiphospholipid syndrome, or history of heparin induced thrombocytopenia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the rate of seroconversion for RVFV neutralizing antibodies 28 days post-vaccination with a single dose of ChAdOx1 RVF | 28 days post-vaccination with one dose of ChAdOx1 RVF
  The proportion of vaccinees in each study group mounting neutralizing antibodies against live RVFV (i.e., seroconversion, as measured by FRNT80

SECONDARY OUTCOMES:
Geometric Mean Antibody Titre for neutralizing antibody titres (GMT) measured by FRNT80 | Days 0, 7, 14, 28, 84, 112, 365 and at 18 months
  Geometric mean antibody titre as measured by FRNT80 for neutralizing antibody titres (GMT) in the single-dose group vs the two-dose group
Geometric mean antibody titre as measured by FRNT80 for IgG antibody titres | Days 0, 7, 14, 28, 84, 112, 365 and at 18 months
  Geometric mean antibody titre as measured by FRNT80 for IgG antibody titres in the single-dose group vs the two-dose group
Spot Forming Units per 1,000,000 PBMCs (SFU/10⁶ PBMCs) for IFN-γ responses to RVFV Gn and Gc glycoproteins measured by enzyme-linked immunospot (ELISpot) assay | Days 0, 7, 14, 28, 84, 112, 365 and at 18 months
  SFU/10⁶ PBMCs for IFN-γ responses to RVFV Gn and Gc glycoproteins measured by enzyme-linked immunospot (ELISpot) assay in the single-dose group vs the two-dose group at Days 0, 7, 14, 28, 84, 112, 365 and at 18 months
T-cells/10^6 PBMCs for multi-functional T cell responses to RVFV Gn and Gc glycoproteins as measured by flow cytometry. | Days 0, 7, 14, 28, 84, 112, 365 and at 18 months.
  T-cells/10^6 PBMCs for multi-functional T cell responses to RVFV Gn and Gc glycoproteins as measured by flow cytometry in the single-dose group vs the two-dose group at Days 0, 7, 14, 28, 84, 112, 365 and at 18 months.
Number of Participants With Serious Adverse Events | Throughout the study, upto 24 months.
  To asses the frequency of serious adverse events (SAEs) throughout the study
Number of participants with solicited, local and systemic adverse events | Day 0-7 and Day 84-91
  frequency of solicited local and systemic adverse events for 7 days following each vaccination.
Number of participants with unsolicited adverse events | throughout the study, upto 24 Months
  Frequency of unsolicited adverse events (AEs) throughout the study
Number of participants with laboratory adverse events | Day 0 and day 28 post vaccination
  Frequency of participants with laboratory adverse events
Number of participants with adverse events of special interest (AESIs) | Throughout the study, upto 24 months
  To asses the frequency of adverse events of special interest (AESIs) throughout the study

OTHER OUTCOMES:
To assess if anti-ChAdOx1 vector immunity influences response to ChAdOx1 RVF vaccination | Day 0 and 84
  Seropositivity rates for anti-ChAdOx1 antibodies as measured by anti-vector neutralizing antibody assay
To estimate exposure to natural RVFV infection in the trial population | Days 0, 28, 84, 112, 365 and at 18 months
  Seropositivity rates for antibodies against RVFV nucleoprotein (antigen not present in ChAdOx1 RVF) as measured by commercial ELISA kit
To assess whether sera from ChAdOx1 RVF vaccinees can passively protect animals from RVFV challenge | Sera collected at day 28 post-vaccination
  Proportion of non-human primates protected from live RVFV challenge following passive immunization with pooled sera from ChAdOx1 RVF vaccinees

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI-Wellcome Trust Research Programme, Kilifi, Coast, Kenya

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be de-identified and coded before sharing.